CLINICAL TRIAL: NCT02796443
Title: When Results of Randomised Controlled Trials and Population Based Studies do Not Reflect the Real World: A Cohort Study in Acute Cholecystitis
Brief Title: The Real World of Acute Cholecystitis
Acronym: REWO
Status: Completed | Type: Observational
Sponsor: Asklepios Klinik Langen (Other)
Collaborators: Goethe University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Ernst Hanisch, Prof. Dr. Dr., Asklepios Klinik Langen
Other Study IDs: AKLangen
Record Dates: First submitted 2016-06-01; First posted 2016-06-10 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Acute Cholecystitis
Keywords: acute cholecystitis; early versus delayed surgery
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Early laparoscopic cholecystectomy (ELC): Operation within 72 hours after onset of symptoms
  Interventions: Procedure: Laparoscopic cholecystectomy (LC)
- Intermediate cholecystectomy (ILC): Operation within 14 days after onset of symptoms
  Interventions: Procedure: Laparoscopic cholecystectomy (LC)
- Delayed LC (DLC): Operation after 6-12 weeks
  Interventions: Procedure: Laparoscopic cholecystectomy (LC)
- Elective laparoscopic cholecystectomy: Biliary colic with no acute cholecystitis
  Interventions: Procedure: Laparoscopic cholecystectomy (LC)

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy (LC) — Removal of the gallbladder via a minimally invasive approach

SUMMARY:
Meta-analysis of randomized controlled trials and population based studies in acute cholecystitis are in favor for early laparoscopic surgery versus a delayed operation several weeks later. The main problems in these studies are the exclusion criteria used, thus not reflecting the real world setting of acute cholecystitis. The purpose of this study is to demonstrate that a delayed laparoscopic cholecystectomy in a real world scenario has no worse outcome in comparison with an early operation (within 72 hours after onset of symptoms).

DETAILED DESCRIPTION:
Background:

Randomized controlled trials (RCTs) and population based studies are in favor of an early operation in acute cholecystitis (1, 2). Thus, one of the largest RCT so far, demonstrated significant more complications in a group of delayed cholecystectomy. The main problems in these studies are the exclusion criteria used, ie severe cases are not considered.

Objective:

In a cohort study all cholecystectomy patients are analysed to demonstrate that delayed laparoscopic cholecystectomy (DLC) in a real world setting has a less complication rate than early cholecystectomy (ELC).

Setting:

Academic Teaching Hospital with 400 beds, seven departments (anesthesiology and intensive care medicine, orthopaedics and trauma surgery, visceral and thoracic surgery, gastroenterology, cardiology, gynecology and obstetrics, psychiatry. The visceral and thoracic department has a main focus on minimally invasive techniques.

Participants:

All cholecystectomy patients during 1/2006 and 9/2015

Variables:

Clavien Dindo Complication score, American Society of Anaesthesiologist (ASA) Score, conversion rate, onset of symptoms, histology, hospital stay

Data sources:

Chart analyses

ELIGIBILITY:
Inclusion Criteria:

* All patients with cholecystectomies

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cholecystectomized patients
Sampling Method: Non-Probability Sample
Enrollment: 1729 (Actual)
Dates: Start 2006-01; Primary Completion 2015-09 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Clavien-Dindo-Complication Score | 3-6 days
  During the hospital stay after Operation, which is usually between 3 and 6 days, all complications according to the Clavien-Dindo-Complication Score, are recorded.

SECONDARY OUTCOMES:
Conversion rate | Intraoperatively
  How often is the laparoscopic approach changed to the open procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ernst W Hanisch, Prof Dr Dr, Principal Investigator — Asklepios Klinik Langen

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be published on www.dkmic.de

REFERENCES:
- [Background] Gutt CN, Encke J, Koninger J, Harnoss JC, Weigand K, Kipfmuller K, Schunter O, Gotze T, Golling MT, Menges M, Klar E, Feilhauer K, Zoller WG, Ridwelski K, Ackmann S, Baron A, Schon MR, Seitz HK, Daniel D, Stremmel W, Buchler MW. Acute cholecystitis: early versus delayed cholecystectomy, a multicenter randomized trial (ACDC study, NCT00447304). Ann Surg. 2013 Sep;258(3):385-93. doi: 10.1097/SLA.0b013e3182a1599b. PMID 24022431
- [Background] de Mestral C, Rotstein OD, Laupacis A, Hoch JS, Zagorski B, Alali AS, Nathens AB. Comparative operative outcomes of early and delayed cholecystectomy for acute cholecystitis: a population-based propensity score analysis. Ann Surg. 2014 Jan;259(1):10-5. doi: 10.1097/SLA.0b013e3182a5cf36. PMID 23979286